CLINICAL TRIAL: NCT07342725
Title: Phase Ib/II Study to Evaluate the Safety and Efficacy of IBI363 in Combination With Chemotherapy as Second-Line Therapy for Unresectable Locally Advanced or Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Principal Investigator, BAIYONG SHEN, professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC-IBI363
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer Metastatic
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Drug: IBI363 + chemotherapy

INTERVENTIONS:
Drug: IBI363 + chemotherapy — IBI363+chemotherapy

SUMMARY:
This study is an Ib/II phase clinical trial evaluating the safety and efficacy of IBI363 combined with chemotherapy as a second-line treatment for unresectable locally advanced or metastatic pancreatic cancer.

Approximately 39-48 patients with unresectable locally advanced or metastatic pancreatic cancer, who have progressed on or are intolerant to first-line chemotherapy (albumin-bound paclitaxel + gemcitabine, AG regimen), will be enrolled. Treatment involves IBI363 combined with chemotherapy and continues until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, or other protocol-specified reasons for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form (ICF)
* Age 18-75 years
* Histologically/cytologically confirmed, unresectable locally advanced or metastatic pancreatic cancer.
* Disease progression or intolerance after first-line treatment with the AG regimen (gemcitabine + albumin-bound paclitaxel).
* ECOG Performance Status(PS) score of 0-1.
* At least one measurable lesion according to RECIST v1.1 criteria.
* Adequate organ and bone marrow function

Exclusion Criteria:

* Previous histologically/cytologically confirmed components including adenosquamous carcinoma, medullary carcinoma, signet ring cell carcinoma, undifferentiated carcinoma, etc.
* Prior treatment with PD-1/PD-L1 inhibitors or other immunotherapies.
* Unresolved > Grade 1 toxicities related to prior anticancer therapy (except persistent Grade 2 alopecia, anemia, peripheral neuropathy, correctable electrolyte abnormalities, or well-controlled endocrine disorders with hormone replacement therapy).
* History of hepatic encephalopathy, seizures, active/new/untreated CNS metastases, spinal compression, carcinomatous meningitis, or leptomeningeal metastases.
* Clinically significant cardiovascular/cerebrovascular diseases
* Known hypersensitivity to IL-2, sintilimab, or monoclonal antibody components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to approximately 36 months
Progression-Free Survival(PFS) | Up to approximately 6 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 6 months
Disease control rate(DCR) | Up to approximately 6 months
Overall Survival(OS) | Up to approximately 12 months